CLINICAL TRIAL: NCT03296397
Title: Efficacy Study of the Quadrivalent Human Papilloma Virus (HPV) Vaccine to Prevent Recurrence of External Genital Warts (EGW) in Patients Who Were Cured in the First Place
Brief Title: Efficacy of Quadrivalent HPV Vaccine to Prevent Relapses of Genital Warts After Initial Therapeutic Response
Acronym: CONDYVAC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P150957
Record Dates: First submitted 2017-07-24; First posted 2017-09-28 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2017-07

CONDITIONS: Genital Warts
Keywords: Genital warts; HPV vaccine; Relapse
MeSH Terms: conditions — Condylomata Acuminata; Recurrence | interventions — Vaccination; Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPV Quadrivalent vaccine (QHV) (Active Comparator): Gardasil
  Interventions: Biological: Vaccination with Gardasil
- Placebo (Placebo Comparator): Normal Saline
  Interventions: Biological: Injection of Normal Saline

INTERVENTIONS:
Biological: Vaccination with Gardasil — Vaccination with Gardasil in patients apparently cured of external genital warts
  Arms: HPV Quadrivalent vaccine (QHV)
Biological: Injection of Normal Saline — Injection of Normal Saline in patients apparently cured of external genital warts
  Arms: Placebo

SUMMARY:
External genital warts (EGW) are a frequent disease (typical yearly incidence of 100 to 200 new cases per 100.000 person-years, typical prevalence of 1 to 4% of the sexually active population), with a heavy toll on patients' quality of life: low self-esteem and severe impairment of sexual well-being are common consequences. Treatments are painful and take time to achieve cure because of low complete remission (20 to 60%) and high recurrence rates (10 to 40%, 30% on average). Finding new means to reduce these recurrence rates thus seems justified. Infection with Human Papillomavirus (HPV) is responsible for EGW,other warts and some epithelial cancers. Out of two currently available HPV vaccines (Cervarix and Gardasil®), only Gardasil® is " quadrivalent " i.e. contains virus like particles imparting protection versus 4 genotypes of HPV, 2 of them responsible of most cancers and pre cancers of the cervix (HPV 16 and 18), and 2 for 90% of EGW (HPV 6 and 11). A close to 100 % efficacy of the quadrivalent HPV vaccine (QHV) on prevention of EGW in naive patients has been shown, leading to their near disappearance in the vaccinated population of countries with a good vaccine coverage. Beside this preventive efficacy, literature data also show that HPV vaccines have an up-to-100% protective effect versus recurrence of destroyed precancerous lesions of the cervix in non-naive patients with an up-to-40 month's follow-up. Also, there is anecdotal evidence that they could help treat severe wart conditions. QHV is also safe and well tolerated when used in a preventive manner.

Investigator hypothesis is that QHV could have a protective effect on the recurrence of EGW in patients who achieve complete remission.

The primary objective is to evaluate if the HPV vaccine, as compared to placebo, reduces the relapse rate of external genital warts over a 12 month-period after their first injection.

The primary endpoint is the Relapse-free "survival". Relapse will have to be clinically confirmed.

The secondary objectives are : 1. To assess the improvement of the quality of life of the patients 2. To investigate the clinical tolerance to three doses of HPV vaccine. The secondary endpoints are

1. Disease relief score as evaluated by patients on a specific questionnaire for Condylomata Acuminata (CECA) and Dermatology Life Quality Index (DLQI) self-administered questionnaires over the treatment and follow-up periods
2. The clinical tolerance to HPV vaccine will be evaluated by assessment of the percentage of patients with local and/or systemic reactions during the study

This is a National multicenter Phase III comparative, double blind randomized, two-parallel groups clinical trial evaluating the efficacy of Gardasil vaccine versus placebo in EGW population. Patients (300) recently cured of EGW will be enrolled over a 18 month-period and will be randomized in a 1:1 ratio to receive three intra muscular (IM) vaccinations of either Gardasil vaccine (150 subjects) or placebo (150 subjects) :

* Group 1: Gardasil (at M0) + Gardasil (at M2) + Gardasil (at M6)
* Group 2: Placebo (at M0) + Placebo (at M2) + Placebo (at M6) Subjects meeting all the inclusion criteria and none of the exclusion criteria will be vaccinated by the investigator or designee of the investigational center and will be examined by the investigator or designee 30 minutes post immunization to assess for local and systemic reactions.

All subjects will be followed by the investigators or designee during the study by phone contacts and visits on site. Diary cards will be used after each vaccination to follow the patients.

Number of visits /participant: 9 Schedule of visits : 1 selection visit (V0) , 3 vaccinations scheduled on site at M0, M2 and M6, 3 phone contacts at M1, M3 and M7, 2 clinical follow up visits on site at M9 and M12 + 1 unscheduled visit on site in case of EGW relapse during the study

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older;
* Patients who, after the nature of the study has been explained to them, and prior to any protocol specific procedures being performed, have given written consent according to local regulatory requirements
* Patients completely cured (no clinically visible lesions) for over two weeks and less than a month prior to inclusion visit (V1, M0) after initial success of classic treatment. If the patient has an EGW relapse, they will not be randomized and will be considered as a screening failure. Screen-failed patients could perform another selection visit after being completely cured (no clinically visible lesions).
* Women of childbearing potential must have a negative pregnancy test and an effective contraception from selection visit (V0) and up to the end of the vaccination period of 6 months;
* Males must have an effective contraception with condoms from selection visit (V0) and up to the end of the vaccination period of 6 months;
* Patients affiliated to a social security regimen;
* Patients able to participate during the 12 months of the study.

Exclusion Criteria:

* Patients with diagnosis of internal ano-genital warts (intra rectal, intra vaginal, intra urethral) at the selection visit
* Patients with positive HIV, Hepatitis C virus (HCV) or Hepatitis B virus (HBV) (Ag HBS) tests;
* Patients whose regular partner(s) have active uncontrolled clinical EGW;
* Patients who received the HPV Vaccine at any time before enrolment to the study;
* Any serious chronic or progressive disease according to the judgement of the investigator;
* Patients with history of an autoimmune disorder or any other known or suspected impairment /alteration of the immune system, or under immunosuppressive therapy including use of systemic corticosteroids or chronic immunosuppressant medication (more than 14 days) (i.e. prednisone, or equivalent ≥10 mg/day) within :

  * the 28 days preceding the first vaccination at the inclusion visit V1 in case of corticosteroids administration
  * the 3 months preceding the first vaccination at the inclusion visit V1 in case of administration of cyclophosphamide, anti-Tumor Necrosis Factor (TNF) alpha , intravenous immunoglobulins, abatacept, corticosteroids as a bolus injection
  * the 6 months preceding the first vaccination at the inclusion visit V1 in case of Cluster of Differentiation antigen 20 (anti-CD20) administration. Topical or inhaled uses of steroid including intranasal are allowed;
* Patients with history of known allergies/hypersensitivity to any component of study vaccine;
* Patients who have any malignancy or lymphoproliferative disorder;
* Patients with thrombocytopenia or coagulation disorder/treatment contra-indicating intramuscular injection;
* Women who are pregnant or are breast-feeding, or are of childbearing age who do not use or do not plan to use acceptable birth control measures, during the first 6 months of the study ;
* Male who do not use or do not plan to use condoms during the first 6 months of the study;
* Patients under a measure of legal protection or unable to consent;
* Patients participating in any clinical trial with another investigational product 28 days prior to first study visit or intent to participate in another clinical study at any time during the conduct of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-11-15 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Relapse free survival (days from first injection) | up to 12 months

SECONDARY OUTCOMES:
Improvement of quality of life by Dermatology Life Quality Index (DLQI) validated scale | at each planned visit/phone contact (1, 2, 3, 6, 7, 9 months), at 12 months (upon end of study visit) or upon premature withdrawal visit
Improvement of quality of life by CECA validated scale | at each planned visit/phone contact (1, 2, 3, 6, 7, 9 months), at 12 months (upon end of study visit) or upon premature withdrawal visit
Clinical tolerance of QHV (percentage of patients with AE) | Day 0
Clinical tolerance of QHV | Month 2 and Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien FOUERE, MD, MSc, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Hôpital St Louis, Paris
  - GH Cochin - Broca - Hôtel-Dieu,, Paris

IPD SHARING:
Plan to Share IPD: Undecided